CLINICAL TRIAL: NCT00854191
Title: A RCT of Mechanical Simulator Practice and Usual Training vs. Usual Training on Novice Trainee Clinical ERCP Performance
Brief Title: Effect of Simulator Practice on Trainees' Endoscopic Retrograde Cholangiopancreatography (ERCP) Performance in the Early Learning Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Joseph Leung, East Bay Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 200804030R
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Patients Undergoing ERCP Examination
Keywords: mechanical simulator; ERCP; training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 4 half-day of simulator ERCP practice and usual training
  Interventions: Device: simulator training
- 2 (Active Comparator): Usual training
  Interventions: Device: simulator training

INTERVENTIONS:
Device: simulator training — 4 half-day of simulator ERCP practice as endoscopist and/or assistant followed by usual training

SUMMARY:
In a RCT, mechanical simulator practice enhances clinical ERCP performance of novice trainees during the first 3 months of usual ERCP training.

DETAILED DESCRIPTION:
Background: The impact of mechanical simulator practice on clinical ERCP performance has not been reported.

Hypothesis: Practice with mechanical simulator improves clinical ERCP performance of novice trainees.

Design: A prospective randomized controlled trial.

Method: 8 trainees without prior ERCP experience from 2 hospitals attended didactic lectures on ERCP. They were randomized in pairs (per hospital) to receive simulator practice and usual training (S) versus usual training only as control (C). Simulator practice included selective bile and pancreatic duct cannulation using a catheter and/or guide wire with different artificial papillae (flat, standard, dual channels) and settings (standard, rotated papilla or duodenum), and exchange of guide wire/accessories and biliary stenting. Local trainers tracked trainees' subsequent clinical ERCP performance for 3 months. Evaluation of trainee skills included success of diagnostic CBD and deep CBD cannulation. Trainer blinded to the randomization provided assessment (1=poor, 5=excellent) of each trainee performed ERCP.

Statistics: Fisher exact test and Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* GI trainees who met the minimum endoscopy training experience

Exclusion Criteria:

* GI trainees with no endoscopy experience

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of trainee skills included success of diagnostic CBD and deep CBD cannulation | 3 months

SECONDARY OUTCOMES:
Trainer blinded to the randomization provided assessment of each trainee performed ERCP | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Liao WC, Leung JW, Wang HP, Chang WH, Chu CH, Lin JT, Wilson RE, Lim BS, Leung FW. Coached practice using ERCP mechanical simulator improves trainees' ERCP performance: a randomized controlled trial. Endoscopy. 2013 Oct;45(10):799-805. doi: 10.1055/s-0033-1344224. Epub 2013 Jul 29. PMID 23897401